CLINICAL TRIAL: NCT00495872
Title: A Multi-Arm Complete Phase 1 Trial of Valproic Acid-Based 2-Agent Oral Regimens for Patients With Advanced Solid Tumor
Brief Title: Valproic Acid-Based 2-Agent Oral Regimens for Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0170
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Advanced Cancer; Dasatinib; Erlotinib; Lapatinib; Lenalidomide; Sorafenib; Erlotinib Hydrochloride; Sunitinib Malate; Sunitinib; Valproic Acid; SU011248
MeSH Terms: interventions — Dasatinib; Erlotinib Hydrochloride; Lapatinib; Lenalidomide; Sorafenib; Sunitinib; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- VN (Experimental): Valproic Acid + Sorafenib
  Interventions: Drug: Sorafenib; Drug: Valproic Acid
- VS (Experimental): Valproic Acid + Sunitinib
  Interventions: Drug: Sunitinib; Drug: Valproic Acid
- VD (Experimental): Valproic Acid + Dasatinib
  Interventions: Drug: Dasatinib; Drug: Valproic Acid
- VT (Experimental): Valproic Acid + Erlotinib
  Interventions: Drug: Erlotinib; Drug: Valproic Acid
- VL (Experimental): Valproic Acid + Lapatinib
  Interventions: Drug: Lapatinib; Drug: Valproic Acid
- VR (Experimental): Valproic Acid + Lenalidomide
  Interventions: Drug: Lenalidomide; Drug: Valproic Acid

INTERVENTIONS:
Drug: Dasatinib — 50 mg by mouth (PO) Twice Daily for 28 Days Every 28 Days
  Other Names: Sprycel®; BMS-354825
  Arms: VD
Drug: Erlotinib — 100 mg PO Daily for 28 Days Every 28 Days
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva
  Arms: VT
Drug: Lapatinib — 1000 mg PO Daily for 28 Days Every 28 Days
  Other Names: GW572016
  Arms: VL
Drug: Lenalidomide — 15 mg PO Daily for 28 Days Every 28 Days
  Other Names: CC-5013; Revlimid™
  Arms: VR
Drug: Sorafenib — 400 mg PO Daily for 21 Days Every 28 Days
  Other Names: BAY 43-9006
  Arms: VN
Drug: Sunitinib — 25 mg PO Daily for 21 Days Every 28 Days
  Other Names: Sunitinib Malate; SU011248
  Arms: VS
Drug: Valproic Acid — 40 mg/kg PO Daily for 7 Days, then 7 Days Off
  Other Names: Depakene

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of valproic acid in combination with either dasatinib, erlotinib hydrochloride, lapatinib, lenalidomide, sorafenib, or SU011248 (sunitinib malate) that can be given to patients with advanced cancer. The safety of each combination of the study drugs will be studied as well.

DETAILED DESCRIPTION:
The Study Drugs:

Valproic acid is designed for use as an anti-seizure medication. It is thought to also have anticancer activity by activating ("turning on") tumor-fighting genes, which may cause cancer cell death.

Dasatinib is designed to change the function of genes. By changing the function of these genes, it may prevent cancer from growing and spreading.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Lapatinib is designed to block the activity of certain molecules. These molecules play a part in the growth of cancer cells and are particularly important for the growth of inflammatory breast cancer tumors.

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Sorafenib is designed to block the function of a cancer protein as well as tumor blood-vessel forming proteins.

Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

Study Administration:

If you are found to be eligible to take part in this study, the study doctor will decide which drug you will receive with valproic acid, based upon your particular disease. You will then begin taking valproic acid plus either dasatinib, erlotinib hydrochloride, lapatinib, lenalidomide, sorafenib, or sunitinib malate. One (1) cycle is either 21 or 28 days long, depending on which study drug combination you receive.

You will take valproic acid by mouth once or twice a day for 7 days in a row. You will then have a 7-day "rest" period from taking this drug.

You will also take either sorafenib or sunitinib malate by mouth once or twice a day continuously for 21 days, or dasatinib, erlotinib hydrochloride, lapatinib, or lenalidomide by mouth once or twice a day continuously for 28 days.

Depending on what stage of the study you are in, you will take the study drugs either once or twice a day.

Study Visits:

You will have the below tests/procedures at designated study visits.

Before each cycle (within 7 days of after your last dose)

* You will be have a complete physical exam.
* Your performance status will be recorded.
* You will be asked about any side effects you may be experiencing.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test. To take part in this study, you must not be pregnant.

After the end of Cycles 2, 4 and 6, you will have a chest x-ray and either a CT scan, MRI scan, or PET scan to check the status of the cancer. You will then have a chest x-ray and either a CT scan, MRI scan, or PET scan after the end of every 3 cycles (Cycle 9, 12, 15, and so on) to check the status of the cancer.

Length of Study:

You will continue to take your study drug combination on this study, as long as the disease does not get worse and you do not experience any intolerable side effects.

End-of-Study Visit:

Once you have stopped taking your study drug combination, you will come back for an end-of-study visit to have the following tests/procedures performed:

* You will have a complete physical exam.
* Your performance status will be recorded.
* Blood may be drawn (about 1 tablespoon) for routine tests
* You may have a CT scan, an MRI scan, or PET to check the status of the cancer, depending on what the study doctor thinks is necessary.

Follow-Up:

The status of the disease will be followed-up for as long as possible after you complete this study. Once every 8 weeks, you will either be contacted by phone and asked how you are feeling (which should take about 5-10 minutes), or you will be asked to come to the clinic for a routine visit. You will have a CT or MRI scan once every 12 weeks (or until another anticancer therapy has been started) to check the status of the cancer.

This is an investigational study. Each of the study drugs is FDA approved and commercially available. The combination of valproic acid plus one of the other study drugs is investigational in this study.

Valproic acid is FDA approved for the treatment of simple and complex absence seizure, complex partial epileptic seizure, acute mania, and migraine prophylaxis.

Dasatinib is FDA approved for the treatment of acute lymphoid leukemia (ALL) and chronic myeloid leukemia (CML).

Erlotinib hydrochloride is FDA approved for the treatment of carcinoma of the pancreas and non-small-cell lung cancer.

Lapatinib is FDA approved for the treatment of breast cancer (inflammatory, relapsed, or refractory) and metastatic breast cancer (HER2 overexpression).

Lenalidomide is FDA approved for the treatment of multiple myeloma and myelodysplastic syndrome.

Sorafenib is FDA approved for the treatment of renal cell carcinoma. Sunitinib malate is FDA approved for the treatment of gastrointestinal stromal tumors and renal cell carcinoma.

Up to 327 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have advanced solid tumor: they have either a disease where there is no established standard of care therapy or have failed one or more prior therapy. (for all treatment arms)
2. Patients must have ECOG performance status < or = 2 (0-2). Patients </=10 years modified Lansky scale >/= 60. Patients >10 to 18 years Karnovsky scale >/= 60.(for all treatment arms)
3. Patients must have normal organ and marrow function as defined below: Platelets > 50,000/uL; Creatinine clearance > 20mL/min (for all treatment arms); Total bilirubin < 5 mg/dL (except for Lapatinib arm); ALT </= 6X ULN for Lapatinib arm only;
4. (cont. from above) Liver function criteria and dosing based on each individual drug: Valproic acid - if ALT >/= 6X ULN or T. Bili >/= 3, then dose should be decreased by 50%; Sorafenib - If Child Pugh class A or B, no dose adjustment; if Child Pugh class C, decrease dose by 50% (400 mg po daily max); Sunitinib - If ALT >/= 6X ULN or T. Bili >/= 3 , decrease dose by 25% (37.5 mg po daily max);
5. (cont. from above) Erlotinib - If ALT > 6X ULN or T. Bili >/= 3 , decrease dose by 25% (100 mg po daily max); Lapatinib - If ALT > 3X ULN or T. Bili > 2X ULN, decrease dose by 60% (500-750 mg po daily max); Dasatinib - No dose adjustment needed; Lenalidomide - No dose adjustment needed.
6. Patients or legal representative must be able to understand and be willing to sign an IRB-approved written informed consent document. (for all treatment arms)
7. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 30 days after the last dose. (for all treatment arms)

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, symptomatic cardiac arrhythmia, active bleeding, active thrombosis, or psychiatric illness/social situations that would limit compliance with study requirements.
2. History of allergic reactions to the study drugs or their analogs.
3. Failure to recover from any prior surgery within 4 weeks of study entry.
4. Any treatment specific for tumor control within 3 weeks of study drugs; or within 2 weeks if cytotoxic agents were given weekly (within 6 weeks for nitrosoureas or mitomycin C), or within 4 half-lives for target agents with half lives and pharmacodynamic effects lasting less than 5 days (that include but are not limited to erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents); or failure to recover from the toxic effect of any therapy prior to study entry.
5. Study agents cannot be obtained for any reason since this study does not provide free agents.
6. Any prior history of hypertensive crisis or hypertensive encephalopathy.
7. Significant vascular disease (e.g., aortic aneurysm, aortic dissection) and symptomatic peripheral vascular disease
8. Evidence of bleeding diathesis or coagulopathy.
9. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
10. Minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
11. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment; and serious, non-healing wound, ulcer, or bone fracture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2007-06; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as Determined by the Number of Participants With Dose Limiting Toxicities | At Day 28 (1 Cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kurzrock R, Atkins J, Wheler J, Fu S, Naing A, Busaidy N, Hong D, Sherman S. Tumor marker and measurement fluctuations may not reflect treatment efficacy in patients with medullary thyroid carcinoma on long-term RET inhibitor therapy. Ann Oncol. 2013 Sep;24(9):2256-61. doi: 10.1093/annonc/mdt177. Epub 2013 May 14. PMID 23676418
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org